CLINICAL TRIAL: NCT04236037
Title: Ultrasound-guided Pleural Biopsy as a Supplement to Thoracentesis: A Randomised Study
Brief Title: Ultrasound-guided Biopsy of the Pleura as a Supplement to Extraction of Fluid in Patients With One-sided Fluid in the Pleura
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It is unrealistic to succeed with sufficient inclusion within the timeframe of the study, why it is terminated.
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-787
Record Dates: First submitted 2019-10-31; First posted 2020-01-22 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Malignant Pleural Effusion; Exudative Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Thoracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided thoracentesis (Active Comparator): Ultrasound guided thoracentesis
  Interventions: Procedure: Thoracentesis
- Ultrasound-guided pleural biopsy and thoracentesis (Experimental): Ultrasound-guided biopsy of the parietal pleura is taken through the same incision as the optimal site for thoracentesis and immediately prior to ultrasound-guided thoracentesis
  Interventions: Procedure: ultrasound-guided pleural biopsy; Procedure: Thoracentesis

INTERVENTIONS:
Procedure: ultrasound-guided pleural biopsy — Using ultrasound the optimal point of entry for thoracentesis is located. Local anesthesia is obtained with 10 mL of 2% lidocaine with adrenalin injected in cutis, subcutis, muscle and pleura. Before removing the syringe, aspiration of pleural fluid confirms the relevance of the chosen site . Again, the area is wiped with disinfectant and a millimeter small skin incision is made with a pointed scalpel. Six US-guided biopsies of 1.2 millimetres using closed needle biopsies (Quick-core Biopsy Needle 18G, COOK Medical, Bloomington, Indiana, USA or Bard Max Core needle 18G, Temple, Arizona, USA). ) are taken from the parietal pleura. Thoracentesis is performed as described above using the same incision as the pleural biopsy.
  Arms: Ultrasound-guided pleural biopsy and thoracentesis
Procedure: Thoracentesis — The optimal point of entry (the largest distance between parietal and visceral pleura) is identified using ultrasound. This is usually on the lower, dorsal side of the chest. Local anesthesia is obtained with 10 mL of 2% lidocaine with adrenalin injected in cutis, subcutis, muscle and pleura. Before removing the syringe, aspiration of pleural fluid confirms the relevance of the chosen site. The area is wiped with disinfectant and a millimeter skin incision is made with a pointed scalpel. A 7 French (or up to 16 French, to the choice of the clinician) pigtail catheter is inserted and connected to sealed bag. Fluid is aspirated via a 3-way valve, and transferred to relevant bottles for culture, analysis of albumin and LDH, protein, and for cytology.

SUMMARY:
The research group will investigate the diagnostic effect of early introduction of ultrasound guided pleural biopsy in the work-up of patients with one-sided pleural effusion, suspected of malignant pleural effusion.

DETAILED DESCRIPTION:
Patients with unilateral pleural effusion with high protein content (exudative pleural effusion) are likely to have malignant pleural effusion. In the Danish guidelines, patient undergo two thoracentesis before more invasive procedures, due to the relatively low incidens of pleural TB and mesothelioma. The aim of the research group is to investigate the effect of early introduction of ultrasound-guided pleural biopsy taken at the optimal sport for thoracentesis. The research group will randomise half of our patients with unilateral pleural exudate to up-front ultrasound-guided biopsy and the other half usual care eg. a second thoracentesis, to see if there is a benefit of early pleural biopsy in the work-up of patients with unilateral pleural effusion, suspected of malignant pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with a previous thoracentesis of a unilateral exudative pleural effusion according to Light's criteria (1) without malignant cells.
* CT thorax or PET-CT with contrast performed.
* Clinical suspicion of cancer such as (but not limited to) weight loss or PET-CT results or former cancer diagnosis.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Bilateral pleural effusions.
* Known cause of pleural effusions.
* Life expectancy <3 months.
* Inability to understand written or spoken Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Proportion of cases with conclusive pleural workup to provide and plan treatment in patients diagnosed with malignant pleural effusion. | 26 weeks post randomization
  Our primary endpoint includes both patients who will receive palliative care and patients who will receive active treatment. For patients receiving palliative care, the presence of malignant cells is sufficient. However, for patients receiving active treatment, the primary endpoint is defined as a definite and treatment-guiding pathological result (immunohistochemistry, mutations, oncodrivers, culture and biochemistry) as decided by a multidisciplinary team conference.

SECONDARY OUTCOMES:
Proportion of cases achieving pleural immunohistochemistry, mutations, oncodrivers and culture. | 26 weeks post randomization
Difference in diagnostic yield between Arm A and Arm B, including subgroup analysis of MPE. | 26 weeks post randomization
Sensitivity of ultrasound-guided closed needle biopsy of parietal pleura for diagnosing malignancy and all causes of PE. | 26 weeks post randomization
Time from inclusion to conclusive, treatment-guiding diagnoses in patients with MPE. | 26 weeks post randomization
The negative likelihood ratio of additional ultrasound-guided closed needle biopsy of parietal pleura in aspect of MPE. | 26 weeks post randomization
Proportion of true non-malignant PE at end of follow-up. | 26 weeks post randomization
Complications to pleural procedures | Day 1 (1 hour after the end of procedure), 7 days and 30 days post-procedure
  mortality, pneumothorax, haemoptysis, local bleeding, infections and hospital admissions
Mean volume pleural fluid drained during thoracentesis | Day 1 within 30 minutes after the end of procedure
  measured in mL
Patient reported discomfort and health | Day 1within 30 minutes after the end of procedure and 7 days post-procedure
  measured by 5Q-5D-5L (2009 EuroQol Group EQ-5D™ Danish version).
Patient reported discomfort and health | Day 1 (immediately before procedure and within 30 minutes after the end of procedure) and 7 days post-procedure
  Measured by Edmonton Symptom Assessment System (ESAS), scale 1-10, 0 being no symptoms, 10 being the worse symptoms
Patient reported cough | Day 1(immediately before procedure and within 30 minutes after the end of procedure) and 7 days post-procedure
  VAS score (visual analogue scale) for cough, 0-10, 0 being no cough, 10 being the worse cough
Pain during procedure | Day 1(within 30 minutes after the end of procedure)
  Measured by VAS score (visual analogue scale) for pain, 0-10, 0 being no pain, 10 being the worse pain
Willingness to repeat the procedure | day og procedure (within 30 minutes after the end of procedure) and 1 week post-procedure
  Measured by 5-point Likert scale,scale 1-5, 1 being definitely willing to have the procedure again, 5 being definitely not willing to have the procedure performed again
Change in patient reported discomfort | Day 1 within 30 minutes after the end of procedure
  iMeasured by Edmonton Symptom Assessment System (ESAS) and VAS score (visual analogue scale) for cough
Changes in patient reported discomfort and health | 7 days post-procedure
  Measured by Edmonton Symptom Assessment System (ESAS) and VAS score (visual analogue scale) for cough and health measured by 5Q-5D-5L (2009 EuroQol Group EQ-5D™ Danish version).
Number of thoracenteses in these 7 days besides the study procedure. | 7 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Bødtger, MD, PhD,, Principal Investigator — Department of Respiratory Medicine; Naestved Hospital, Denmark
Locations (2):
- Denmark (2):
  - Næstved Sygehus, department of pulmonary medicine, Næstved, Region Sjælland
  - Zealand University Hospital, Roskilde, Department of Pulmonary medicine, Roskilde, Region Sjælland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Light RW, Macgregor MI, Luchsinger PC, Ball WC Jr. Pleural effusions: the diagnostic separation of transudates and exudates. Ann Intern Med. 1972 Oct;77(4):507-13. doi: 10.7326/0003-4819-77-4-507. No abstract available. PMID 4642731